CLINICAL TRIAL: NCT06534983
Title: A Randomized Phase II, Double-blind, Multicenter Study Evaluating the Efficacy and Safety of Autogene Cevumeran Plus Nivolumab Versus Nivolumab as Adjuvant Therapy in Patients With High-risk Muscle-invasive Urothelial Carcinoma
Brief Title: A Study to Evaluate the Efficacy and Safety of Autogene Cevumeran With Nivolumab Versus Nivolumab Alone in Participants With High-risk Muscle-invasive Urothelial Carcinoma (MIUC)
Acronym: IMCODE004
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO45230; 2023-509023-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Muscle-invasive Urothelial Carcinoma
MeSH Terms: interventions — Nivolumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Autogene Cevumeran + Nivolumab (Experimental): Participants will receive autogene cevumeran along with nivolumab intravenously (IV) at a recommended dose at specified timepoints.
  Interventions: Drug: Autogene Cevumeran; Drug: Nivolumab
- Saline + Nivolumab (Active Comparator): Participants will receive saline solution along with 480 milligrams (mg) of nivolumab, IV, once every 4 weeks (Q4W) for 1 year.
  Interventions: Drug: Nivolumab; Drug: Saline

INTERVENTIONS:
Drug: Autogene Cevumeran — Autogene cevumeran will be administered as an IV infusion per the schedule specified in the arm.
  Other Names: RO7198457
  Arms: Autogene Cevumeran + Nivolumab
Drug: Nivolumab — Nivolumab will be administered as an IV infusion per the schedule specified in the arm.
  Other Names: Opdivo
Drug: Saline — Saline solution for IV infusion.
  Arms: Saline + Nivolumab

SUMMARY:
The main purpose of the study is to evaluate the efficacy of adjuvant treatment with autogene cevumeran plus nivolumab compared with nivolumab in participants with high risk MIUC.

In this study participants will be enrolled in a safety run-in phase to receive autogene cevumeran + nivolumab. This phase will be conducted to monitor and ensure the safety of study participants. After all participants in the safety run-in have been enrolled to receive autogene cevumeran + nivolumab, further participants will be randomized in either autogene cevumeran + nivolumab or the saline + nivolumab arm.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have the capacity to participate/enroll in the study and to provide informed consent
* Histologically confirmed muscle-invasive UC (also termed transitional cell carcinoma [TCC]) of the bladder or upper urinary tract
* Tumor-node-metastasis (TNM ) classification (Union for International Cancer Control [UICC]/American Joint Committee on Cancer [AJCC] 7th edition) at pathological examination of surgical resection specimen of (y)pT3-4 or (y)pN+ and M0
* Surgical resection of MIUC of the bladder or upper tract
* Participants who have received neoadjuvant chemotherapy (NAC), including antibody drug-conjugate, either alone or in combination with a checkpoint inhibitor (CPI), are eligible
* Participants who have not received any prior NAC are also eligible, provided they meet one of the following criteria, which would make them ineligible to receive adjuvant cisplatin-based therapy: participant refusal, cisplatin ineligibility or investigator decision
* Tumor tissue must be provided for biomarker analysis
* Absence of residual disease and absence of metastasis, as confirmed by a negative baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan of the pelvis, abdomen, and chest no more than 28 days prior to randomization
* Full recovery from cystectomy or nephroureterectomy within 120 days following surgery
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Negative human immunodeficiency virus (HIV) test at screening
* Negative hepatitis B surface antigen (HbsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb), or a negative HBsAb at screening accompanied by either of the following: negative total hepatitis B core antibody (HBcAb) or positive total HBcAb test followed by quantitative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) < 500 international units/milliliter (IU/mL)
* Negative hepatitis C virus (HCV) antibody test at screening, or a positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening

Exclusion Criteria:

* Partial cystectomy in the setting of bladder cancer primary tumor or partial nephroureterectomy in the setting of renal pelvis primary tumor
* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment
* Adjuvant chemotherapy, immunotherapy, or radiation therapy for UC following surgical resection
* Prior active malignancies within 3 years prior to randomization
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2029-03-07 (Estimated); Study Completion 2034-01-06 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed (INV) Disease-free Survival (DFS) | Randomization until the first recurrence of disease or death from any cause, whichever occurs first (approximately 6 years)
  Disease recurrence is defined as any of the following:
  * Local (pelvic) recurrence of urothelial carcinoma (UC) (including soft tissue and regional lymph nodes);
  * Urinary tract recurrence of UC (excluding low-grade non-muscle-invasive bladder cancer [NMIBC]);
  * Distant metastasis of UC.

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization until the date of death from any cause (approximately 6 years)
INV-DFS in Programmed Death Ligand-1 (PD-L1) Expression ≥ 1% Population | Randomization until first occurrence of a documented disease recurrence or death from any cause, whichever occurs first (approximately 6 years)
INV-Distant Metastasis-free Survival (DMFS) | Randomization to the date of diagnosis of distant (i.e., non-locoregional) metastases (approximately 6 years)
Number of Participants With Adverse Events (AEs) | Up to approximately 22 months
Change From Baseline in Participant-reported Pain, Physical Function, Role Function and Quality of Life (QoL) as Assessed Using European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire-C30 (EORTC QLQ-C30) | From Day 1 up to approximately 25 months
  The EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning scale, three symptom scales, global health status (GHS), QoL, and single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Scale scores can be obtained for the multi-item scales. The functioning and symptoms items are scored on a 4-point scale that ranges from "not at all" to "very much", and the GHS and QoL items are scored on a 7-point scale that ranges from "very poor" to "excellent". Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of functioning/QoL.
Number of Participants With Symptomatic Treatment Toxicities as Assessed by National Cancer Institute Patient-reported Outcomes - Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) | From Day 1 up to Cycle 21 (cycle length=28 days)
  The PRO-CTCAE contains 124 questions that are rated either dichotomously (for determination of presence vs. absence) or on a 5-point Likert scale (for determination of frequency of occurrence, severity, and interference with daily function). Treatment toxicities can occur with observable signs (e.g., vomiting) or non-observable symptoms (e.g., nausea). A subset of 16 symptoms (fatigue, chills, nausea, vomiting, diarrhea, constipation, decreased appetite, swelling, itching, rash, headache, muscle pain, joint pain, general pain, cough, and shortness of breath) will be assessed.
Number of Participants Experiencing AE Burden due to Treatment as Assessed by EORTC Item Library 46 (IL46) | From Day 8 up to Cycle 21 (cycle length=28 days)
  The EORTC IL46 is a single question that assesses bother (burden) of treatment. It is rated on a scale from 1 to 4, ranging from "not at all" to "very much".
Change from Baseline in Symptomatic Treatment Toxicities as Assessed by NCI PRO-CTCAE | From Day 1 up to Cycle 21 (cycle length=28 days)
  The PRO-CTCAE contains 124 questions that are rated either dichotomously (for determination of presence vs. absence) or on a 5-point Likert scale (0=none to 4=very much) for determination of frequency of occurrence, severity, and interference with daily function. Treatment toxicities can occur with observable signs (e.g., vomiting) or non-observable symptoms (e.g., nausea). A subset of 16 symptoms (fatigue, chills, nausea, vomiting, diarrhea, constipation, decreased appetite, swelling, itching, rash, headache, muscle pain, joint pain, general pain, cough, and shortness of breath) will be assessed in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (105):
- United States (26):
  - Highlands Oncology Group., Springdale, Arkansas
  - Kaiser Permanente - Baldwin Park, Baldwin Park, California
  - City of Hope Cancer Center, Duarte, California
  - Kaiser Permanente - Los Angeles (N. Vermont), Los Angeles, California
  - Kaiser Permanente - Riverside, Riverside, California
  - University of California San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Norton Cancer Institute, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSK Nassau, Uniondale, New York
  - Providence Portland Medical Ctr, Portland, Oregon
  - AHN Cancer Institute ? Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Bon Secours - St. Francis Hospital, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Argentina (3):
  - Instituto Alexander Fleming, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Hospital Italiano, Ciudad Autonoma Buenos Aires
- Australia (3):
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Belgium (4):
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Ste-Elisabeth, Namur
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Herlev Hospital, Herlev
- France (4):
  - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Vivantes Klinikum Am Urban, Berlin
  - Universitätsklinikum Düsseldorf;Urologische Klinik, Düsseldorf
  - Uniklinik Essen, Essen
  - Uniklinik-Eppendorf, Hamburg
  - Uniklinikum Heidelberg, Heidelberg
  - Marien Hospital Herne, Herne
  - Universitätsklinikum Jena, Urologische Klinik und Poliklinik, Jena
  - Klinikum rechts der Isar der TU München, München
  - Klinikum Stuttgart - Katharinenhospital, Stuttgart
  - Universitätsklinikum Ulm, Ulm
- Greece (3):
  - Alexandras Hospital, Athens
  - Attikon University General Hospital, Athens
  - Theageneio Hospital, Thessaloniki
- Italy (9):
  - A.O. Universitaria Ospedale Consorziale Policlinico Di Bari, Bari, Apulia
  - Istituto Nazionale Tumori Irccs Fondazione G. Pascale, Napoli, Campania
  - AZ.Osp S. Orsola ? Malpighi-Reparto di Oncologia Medica, Bologna, Emilia-Romagna
  - IFO - Istituto Regina Elena, Rome, Lazio
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - A.O. Universitaria S. Luigi Gonzaga, Orbassano, Piedmont
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
  - A.O.U di Verona Policlinico G.B. Rossi, Verona, Veneto
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - St. Antonius locatie Leidsche Rijn, Utrecht
- Akershus universitetssykehus, Lørenskog, Norway
- Poland (7):
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - Szpital Wojewodzki im. M. Kopernika w Koszalinie, Koszalin
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli, Lublin
  - Szpital Kliniczny Ministerstwa Spraw Wewn?trznych i Administracji z Warmi?sko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Radomskie Centrum Onkologii, Radom
  - AIDPORT Sp. z o. o., Skórzewo
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Sant Andreu de la Barca, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano Oncologia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes Onkologiska Klinik, Universitetssjukhuset, Lund
- Taiwan (3):
  - Chang Gung Medical Foundation - Kaohsiung, Kaohsiung City
  - National Taiwan Uni Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Clatterbridge Cancer Centre, Bebington
  - Royal Devon and Exeter Hospital, Exeter
  - Barts & London School of Med;Medical Oncology, London
  - Royal Preston Hosptial, Preston
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing